CLINICAL TRIAL: NCT03472872
Title: A Randomized Double-blind Comparative Efficacy Trial of IV Acetaminophen Versus IV Ketorolac for Emergency Department Treatment of Generalized Headache
Brief Title: A Comparative Efficacy Trial of IV Acetaminophen Versus IV Ketorolac for Emergency Department Treatment of Generalized Headache
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no longer recruiting or studying
Sponsor: Corewell Health South (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMMC#1569
Record Dates: First submitted 2018-02-26; First posted 2018-03-21 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Headache
Keywords: acetaminophen; ketorolac; prochlorperazine; diphenhydramine
MeSH Terms: conditions — Headache | interventions — Ketorolac; Ketorolac Tromethamine; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind trial comparing two parenteral adjuvant treatments for headache among patients presenting to the Lakeland Health Emergency Department in St. Joseph, MI.
Who Masked: Participant, Care Provider
Masking Description: The provider will place orders in the electronic medical record for "Headache study order set". This order set includes Compazine® 10 mg IV, Benadryl® 25 mg IV, and "study drug". Pharmacy will receive the order for the study drug. The research pharmacist will randomly assign participants to group A (1000 mg Ofirmev®) or group B (15 mg ketorolac).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac Arm (Experimental): The patient will receive a 0.9% normal saline bolus of 1,000ml at 500ml/hr, 25mg diphenhydramine IV, 10mg prochlorperazine IV, 15mg ketorolac in 100mL 0.9% normal saline IVPB
  Interventions: Drug: Ketorolac
- Acetaminophen Arm (Experimental): The patient will receive a 0.9% normal saline bolus of 1,000ml at 500ml/hr, 25mg diphenhydramine IV, 10mg prochlorperazine IV, 1,000mg acetaminophen in a 100ml IVPB
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Ketorolac — 15mg ketorolac in 100mL 0.9% normal saline IVPB 1,000mg acetaminophen in a 100ml IVPB
  Other Names: Toradol
  Arms: Ketorolac Arm
Drug: Acetaminophen — 1,000mg acetaminophen IVPB
  Other Names: Ofirmev
  Arms: Acetaminophen Arm

SUMMARY:
This randomized, double-blind trial will compare the clinical efficacy of IV acetaminophen to that of IV ketorolac as adjuncts to standard therapy (prochlorperazine and diphenhydramine) in the treatment of patients presenting to the emergency department with chief complaint of "headache" or variants thereof.

DETAILED DESCRIPTION:
After initial assessment of the patient by the provider, including careful review of inclusion and exclusion criteria, informed consent will be obtained. If a patient does not wish to participate in this study, he/she will receive alternative treatment at the discretion of their ED provider.

The provider will place orders in the electronic medical record for "Headache study order set". This order set includes Compazine® 10 mg IV, Benadryl® 25 mg IV, and "study drug". Pharmacy will receive the order for the study drug. The research pharmacist will randomly assign participants to group A (1000 mg Ofirmev®) or group B (15 mg ketorolac). He/she will fill medication vials and IV bags in each "study kit". The kit for group A will contain a 100mL bag containing 1000 mg acetaminophen and a placebo vial of normal saline as well as both Compazine® and Benadryl®. The kit for group B will contain 100mL 0.9% normal saline and a vial containing 15 mg ketorolac as well as Compazine® and Benadryl®. The "study kit" will be sent to the emergency department via the tube system. When the study kit arrives, he/she will give each patient Compazine® and Benadryl®, hang the IV bag, and administer the contents of the vial. Therefore, every patient will receive a "push" of the contents in the vial (ketorolac or normal saline) and an 100mL infusion (Ofirmev or normal saline).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Presenting chief complaint of headache, migraine, tension headache, cluster headache, or headache not otherwise specified
* Report of pain 4 using a standard 11-point numerical scale (0 to 10; 0=no pain and 10=worst possible pain)

Exclusion Criteria:

* Age < 18 years or > 65 years
* Inability to provide informed consent
* Physical or mental disability hindering adequate response to assessment of pain
* Hemodynamic instability/medical condition requiring acute life-saving medical intervention
* Documented or suspected pregnancy or currently breastfeeding
* Known brain mass, intracranial hemorrhage, skull fracture
* Known allergy, hypersensitivity, or prior adverse reaction to acetaminophen, NSAIDs, diphenhydramine, or prochlorperazine
* Known contraindications to acetaminophen use

  * Severe hepatic impairment, severe active liver disease
* Known contraindications to ketorolac/NSAID use

  * Active bleeding, peptic ulcer disease, bleeding dyscrasias
* Known contraindication to diphenhydramine use
* Known contraindication to prochlorperazine use

  * Comatose states or in the presence of large amounts of CNS depressants
* Patients who have consumed

  * > 2600 mg acetaminophen within the past 24 hours
  * > 500 mg acetaminophen within the previous 4 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-06-14 (Actual)

PRIMARY OUTCOMES:
Pain Improvement | 60 minutes
  Comparison of the improvement in pain score between baseline and 60 minutes following analgesic administration, assessed using a Numeric Pain Rating Scale ( RATE PAIN FROM 0-10, with 0 = no pain and 10 = worst possible pain)

SECONDARY OUTCOMES:
pain score at 30 minutes | 30 minutes
  ED staff will re-assess the patient and record level of pain at time of study drug administration and at 30 minutes after study drug administration, pain assessed using a Numeric Pain Rating Scale ( RATE PAIN FROM 0-10, with 0 = no pain and 10 = worst possible pain)
pain score at 90 minutes | 90 minutes
  ED staff will re-assess the patient and record level of pain at time of study drug administration and at 90 minutes after study drug administration, pain assessed using a Numeric Pain Rating Scale ( RATE PAIN FROM 0-10, with 0 = no pain and 10 = worst possible pain)
need for rescue medication in the ED | 90 minutes
  ED staff will re-assess the patient and record level of pain at time of study drug administration and at 90 minutes after study drug administration, pain assessed using a Numeric Pain Rating Scale ( RATE PAIN FROM 0-10, with 0 = no pain and 10 = worst possible pain)
patient's desire to receive the same medication again | 90 minutes
  prior to discharge the ED staff will ask the patient if they would like to receive the same medication again.
Need for rescue medication | 90 minutes
  If a rescue medication is required, the time, pain level, and type of medication given will be recorded. pain assessed using a Numeric Pain Rating Scale ( RATE PAIN FROM 0-10, with 0 = no pain and 10 = worst possible pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Lakeland Regional Healthcare, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burch RC, Loder S, Loder E, Smitherman TA. The prevalence and burden of migraine and severe headache in the United States: updated statistics from government health surveillance studies. Headache. 2015 Jan;55(1):21-34. doi: 10.1111/head.12482. Erratum In: Headache. 2015 Feb;55(2):356. PMID 25600719
- [Background] Derry S, Moore RA. Paracetamol (acetaminophen) with or without an antiemetic for acute migraine headaches in adults. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD008040. doi: 10.1002/14651858.CD008040.pub3. PMID 23633349
- [Background] Gungor F, Akyol KC, Kesapli M, Celik A, Karaca A, Bozdemir MN, Eken C. Intravenous dexketoprofen vs placebo for migraine attack in the emergency department: A randomized, placebo-controlled trial. Cephalalgia. 2016 Feb;36(2):179-84. doi: 10.1177/0333102415584604. Epub 2015 May 5. PMID 25944813
- [Background] Florence CS, Zhou C, Luo F, Xu L. The Economic Burden of Prescription Opioid Overdose, Abuse, and Dependence in the United States, 2013. Med Care. 2016 Oct;54(10):901-6. doi: 10.1097/MLR.0000000000000625. PMID 27623005
- [Background] Friedman BW, Cabral L, Adewunmi V, Solorzano C, Esses D, Bijur PE, Gallagher EJ. Diphenhydramine as Adjuvant Therapy for Acute Migraine: An Emergency Department-Based Randomized Clinical Trial. Ann Emerg Med. 2016 Jan;67(1):32-39.e3. doi: 10.1016/j.annemergmed.2015.07.495. Epub 2015 Aug 29. PMID 26320523
- [Background] Friedman BW, Adewunmi V, Campbell C, Solorzano C, Esses D, Bijur PE, Gallagher EJ. A randomized trial of intravenous ketorolac versus intravenous metoclopramide plus diphenhydramine for tension-type and all nonmigraine, noncluster recurrent headaches. Ann Emerg Med. 2013 Oct;62(4):311-318.e4. doi: 10.1016/j.annemergmed.2013.03.017. Epub 2013 Apr 6. PMID 23567060
- [Background] Friedman BW, Esses D, Solorzano C, Dua N, Greenwald P, Radulescu R, Chang E, Hochberg M, Campbell C, Aghera A, Valentin T, Paternoster J, Bijur P, Lipton RB, Gallagher EJ. A randomized controlled trial of prochlorperazine versus metoclopramide for treatment of acute migraine. Ann Emerg Med. 2008 Oct;52(4):399-406. doi: 10.1016/j.annemergmed.2007.09.027. Epub 2007 Nov 19. PMID 18006188
- [Background] Friedman BW, West J, Vinson DR, Minen MT, Restivo A, Gallagher EJ. Current management of migraine in US emergency departments: an analysis of the National Hospital Ambulatory Medical Care Survey. Cephalalgia. 2015 Apr;35(4):301-9. doi: 10.1177/0333102414539055. Epub 2014 Jun 19. PMID 24948146
- [Background] Jones J, Sklar D, Dougherty J, White W. Randomized double-blind trial of intravenous prochlorperazine for the treatment of acute headache. JAMA. 1989 Feb 24;261(8):1174-6. PMID 2915441
- [Background] Lipton RB, Baggish JS, Stewart WF, Codispoti JR, Fu M. Efficacy and safety of acetaminophen in the treatment of migraine: results of a randomized, double-blind, placebo-controlled, population-based study. Arch Intern Med. 2000 Dec 11-25;160(22):3486-92. doi: 10.1001/archinte.160.22.3486. PMID 11112243
- [Background] Lucado J, Paez K, Elixhauser A. Headaches in U.S. Hospitals and Emergency Departments, 2008. 2011 May. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #111. Available from http://www.ncbi.nlm.nih.gov/books/NBK56047/ PMID 21735579
- [Background] Bukharin OV, Tolstov IuP, Anikin IA. [Indices of natural nonspecific immunity in chronic tonsillitis]. Vestn Otorinolaringol. 1975 Jan-Feb;(1):61-4. No abstract available. Russian. PMID 1114616
- [Background] Masoumi K, Forouzan A, Asgari Darian A, Feli M, Barzegari H, Khavanin A. Comparison of clinical efficacy of intravenous acetaminophen with intravenous morphine in acute renal colic: a randomized, double-blind, controlled trial. Emerg Med Int. 2014;2014:571326. doi: 10.1155/2014/571326. Epub 2014 Aug 13. PMID 25197573
- [Background] Needleman SM. Safety of rapid intravenous of infusion acetaminophen. Proc (Bayl Univ Med Cent). 2013 Jul;26(3):235-8. doi: 10.1080/08998280.2013.11928969. PMID 23814378
- [Background] Orr SL, Friedman BW, Christie S, Minen MT, Bamford C, Kelley NE, Tepper D. Management of Adults With Acute Migraine in the Emergency Department: The American Headache Society Evidence Assessment of Parenteral Pharmacotherapies. Headache. 2016 Jun;56(6):911-40. doi: 10.1111/head.12835. PMID 27300483
- [Background] Pardutz A, Schoenen J. NSAIDs in the Acute Treatment of Migraine: A Review of Clinical and Experimental Data. Pharmaceuticals (Basel). 2010 Jun 17;3(6):1966-1987. doi: 10.3390/ph3061966. PMID 27713337
- [Background] Shrestha M, Singh R, Moreden J, Hayes JE. Ketorolac vs chlorpromazine in the treatment of acute migraine without aura. A prospective, randomized, double-blind trial. Arch Intern Med. 1996 Aug 12-26;156(15):1725-8. PMID 8694672
- [Background] Taggart E, Doran S, Kokotillo A, Campbell S, Villa-Roel C, Rowe BH. Ketorolac in the treatment of acute migraine: a systematic review. Headache. 2013 Feb;53(2):277-87. doi: 10.1111/head.12009. Epub 2013 Jan 8. PMID 23298250
- [Background] Turkcuer I, Serinken M, Eken C, Yilmaz A, Akdag O, Uyan E, Kiray C, Elicabuk H. Intravenous paracetamol versus dexketoprofen in acute migraine attack in the emergency department: a randomised clinical trial. Emerg Med J. 2014 Mar;31(3):182-5. doi: 10.1136/emermed-2013-203044. Epub 2014 Jan 6. PMID 24394884
- [Background] Vinson DR, Drotts DL. Diphenhydramine for the prevention of akathisia induced by prochlorperazine: a randomized, controlled trial. Ann Emerg Med. 2001 Feb;37(2):125-31. doi: 10.1067/mem.2001.113032. PMID 11174228
- [Background] Vinson DR, Hurtado TR, Vandenberg JT, Banwart L. Variations among emergency departments in the treatment of benign headache. Ann Emerg Med. 2003 Jan;41(1):90-7. doi: 10.1067/mem.2003.24. PMID 12514688
- See also: Related Info — http://www.accessdata.fda.gov/drugsatfda_docs/label/2005/010571s096lbl.pdf
- See also: Related Info — http://www.accessdata.fda.gov/drugsatfda_docs/label/2010/022450lbl.pdf
- See also: Related Info — http://www.accessdata.fda.gov/drugsatfda_docs/label/2013/019645s019lbl.pdf
- See also: Related Info — http://www.accessdata.fda.gov/drugsatfda_docs/label/2013/091526lbl.pdf